CLINICAL TRIAL: NCT04429113
Title: Is the Quad Helix More Efficient to Correct Mandibular Asymmetry Before Age 7? A Retrospective Comparative Study
Brief Title: Quad Helix and Correction of Mandibular Asymmetry
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0350
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Mandibular Asymmetry; Functional Shift of the Mandible
Keywords: Early treatment; Posterior unilateral cross bite; Quad helix
MeSH Terms: interventions — Palatal Expansion Technique

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- G1 or Early Group: Patients treated before age 7 (Quad Helix on decidual second molars)
  Interventions: Device: Maxillary expansion with conventional Quad Helix bonded on molars.
- G2 or Late Group: Patients treated between 7 and 13 years old (Quad Helix on first permanent molars)
  Interventions: Device: Maxillary expansion with conventional Quad Helix bonded on molars.

INTERVENTIONS:
Device: Maxillary expansion with conventional Quad Helix bonded on molars. — Maxillary expansion with conventional Quad Helix bonded on molars

SUMMARY:
To compare the effectiveness of the Quad Helix, an orthopaedic conventional appliance, in the correction of skeletal mandibular asymmetry, on frontal x-ray, in subjects treated before or after 7 years.

DETAILED DESCRIPTION:
Introduction : Unilateral posterior crossbite (UPCB), often from dysfunctional and para-functional causes, leads to positional mandibular asymmetries that can develop at a very young age into skeletal mandibular deviation; hence the interest of early maxillary expansion. The purpose of this retrospective study was to compare the impact of maxillary expansion by Quad Helix (QH) on mandibular skeletal asymmetry correction before and after 7 years of age.

Materials and methods : All children with UPCB and skeletal mandibular asymmetry, who were treated by QH in the orthodontic department between February 2017 and August 2018 and who have done a radiography file at baseline (T0) and 12 months later (T1) have been included. The patients were divided into two groups according to age: under 7 years of age (early group G1) with QH adjusted on second primary molars and over up to 13 years old (late group G2) with QH adjusted on first permanent molars. The differences between the right and left sides of the mandible in corpus length L (main eligibility criterion) and ramus height H (secondary criterion) were compared between groups. X² test, Fisher's exact test and Wilcoxon rank-sum tests were used for baseline comparisons. A multifactorial analysis allowing adjustment on possible confounding factors was used with R software at a significance level of 5%.

ELIGIBILITY:
Inclusion criteria:

* Unilateral Posterior Crossbite (at least one tooth) and skeletal mandibular asymmetry
* Treated by Quad Helix in the Orthodontic Department of the CHU Montpellier
* with frontal X-rays available at baseline and 12months later

Exclusion criteria:

* Incomplete File
* Inadequate quality of x-rays

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients of Orthodontic Department of the CHU of Montpellier
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Difference in the mandibular corpus length between the right and left side | 1 day
  Difference in the mandibular corpus length between the right and left side : △L on conventional frontal x-ray.

SECONDARY OUTCOMES:
Difference in the mandibular ramus height between the right and left side of the mandibule | 1 day
  Difference in the mandibular ramus height between the right and left side of the mandibule : △H on conventional frontal x-ray.

CONTACTS AND LOCATIONS:
Overall Officials: Manon Fourneron, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC